CLINICAL TRIAL: NCT06491199
Title: HABPY: Home Assessment of Blood Pressure in PregnancY
Brief Title: Home Assessment of Blood Pressure in PregnancY
Acronym: HABPY
Status: Not yet recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Women's Health Research Institute of British Columbia (Other); Providence Healthcare (Other); Fraser Health (Other)
Responsible Party: Principal Investigator, Karen Tran, Clinical Assistant Professor, General Internal Medicine, University of British Columbia
Other Study IDs: H23-03815
Record Dates: First submitted 2024-06-11; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Hypertensive Disorder of Pregnancy
MeSH Terms: conditions — Toxemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Home blood pressure telemonitoring program and clinician monitoring — Home Blood Pressure Telemonitoring (HBPT) includes used of an app to collect and transmit blood pressure readings.
  Clinician monitoring includes OBIM physicians reviewing transmitted BP data and contacting patients to adjust antihypertensive medication regimens.

SUMMARY:
The goal of this observational study is to evaluate the feasibility and safety of a comprehensive home blood pressure telemonitoring (HBPT) program for pregnant people with hypertensive disorders of pregnancy (HDP).

Participants will receive training on the use of a home BP telemonitor with tele-transmission function for the remainder of their pregnancy and 6 weeks postpartum. Participating obstetric internal medicine (OBIM) clinicians will monitor the transmitted values and adjust anti-hypertensive medications based on the home BP readings.

Our primary goal is to describe the feasibility and safety of a comprehensive HBPT pilot program in British Columbia, Canada (BC).

Secondary research questions will address:

1. What is the end-user acceptability of a comprehensive HBPT pilot program in BC?
2. What are the effects of a comprehensive HBPT pilot program on factors such as:

1. Maternal and neonatal outcomes 2. Home blood pressure (BP) metrics 3. Process measures 4. Anti-hypertensive medications 5. Fidelity to interventions 6. Health Care utilization

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥ 19 years
* Pregnancy
* Gestational age 20+0 to 36+0 weeks gestational age
* Diagnosed with gestational hypertension (defined as SBP ≥140 mm Hg and/or DBP ≥ 90 mm Hg) after 20 weeks gestation OR Chronic hypertension (defined as SBP ≥140 mm Hg and/or DBP ≥ 90 mm Hg), present at booking or before 20 weeks gestation, or receiving treatment (including lifestyle measures) prior to pregnancy and/or at time of referral OR Transient elevated office BP reading (defined as one time reading of SBP ≥140 mm Hg and/or DBP ≥ 90 mm Hg with risk factors for HDP as per Canadian guidelines).
* Participant is willing and able to give informed consent for participation in the study
* Able and willing to comply with study requirements
* Has smart phone

Exclusion Criteria:

* Anticipated inpatient admission
* Remaining pregnancy less than 2 weeks duration
* Imminent delivery (within the next 48 hours)
* Non-English speaking or no family members who can help translate

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who are pregnant between 20+0 weeks and 26+0 weeks diagnosed with a hypertensive disorder of pregnancy (HDP) such as chronic hypertension, gestational hypertension, or transient elevated blood pressure with HDP risk factors.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility: recruitment rate of HBPT program | From time of enrolment to 6 weeks post partum
  Average number of participants who are screened and eligible who consent to participate in this study per month of recruitment.
Feasibility: retention rate of HBPT program | From time of enrolment to 6 weeks post-partum
  Rate of patients who are consented and enrolled in study and participate for the duration of the study period compared to those who are lost to follow-up or attrite during the study period.
Safety: Proportion of participants with severe hypertension. | From time of enrolment to 6 weeks post-partum
  Number of patients who experience severe hypertension (defined as office/obstetrical visits/home systolic blood pressure (SBP) ≥ 160 mm Hg and/or diastolic blood pressure (DBP) ≥ 110 mm Hg) as a proportion of total study population.
Safety: Incidence density of study participants with severe hypertension | From time of enrolment to 6 weeks post-partum.
  Proportion of new cases of severe hypertension (defined as office/obstetrical visits/home systolic blood pressure (SBP) ≥ 160 mm Hg and/or diastolic blood pressure (DBP) ≥ 110 mm Hg) divided by the total person-time from enrolment to 6 weeks post-partum.

SECONDARY OUTCOMES:
End-user acceptability of comprehensive HBPT program based on EuroQol 5 Dimension 5 Level | From time of enrolment to end of study period (6 weeks postpartum).
  The EuroQol-5D-5L survey is a standardized instrument used to measure health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each with five levels of severity, 1 being the least severe and 5 being the most severe. Acceptability based on change in score from enrolment to end of study period.
End-user acceptability of comprehensive HBPT program based on Spielberger State-Trait Anxiety Inventory 6 (STAI-6) questionnaire. | From time of enrolment to end of study period (6 weeks postpartum).
  Health-related quality of life will be assessed by EuroQol 5 Dimension 5 Level (EQ-5D-5L) questionnaire; Anxiety will be assessed based on Spielberger State-Trait Anxiety Inventory 6 The State-Trait Anxiety Inventory (STAI) survey is a psychological assessment tool used to measure both temporary (state) and long-standing (trait) levels of anxiety in individuals. he State-Trait Anxiety Inventory (STAI) consists of two subscales: the State Anxiety (S-Anxiety) scale and the Trait Anxiety (T-Anxiety) scale, each with 20 items.
  Minimum value: 20 (for each subscale) Maximum value: 80 (for each subscale) Interpretation of scores: Higher scores indicate higher levels of anxiety, meaning a worse outcome in terms of anxiety levels. Acceptability based on change in score from enrolment to end of study period.
End-user acceptability of comprehensive HBPT program based on Patient Satisfaction Questionnaire Short Form (PSQ-18). | From time of enrolment to end of study period (6 weeks postpartum).
  xconcise survey designed to measure patient satisfaction across multiple dimensions of healthcare, including technical quality, interpersonal manner, communication, and financial aspects.
  Patient Satisfaction Questionnaire Short Form survey designed to measure patient satisfaction across multiple dimensions of healthcare, including technical quality, interpersonal manner, communication, and financial aspects. Acceptability based on change in score from enrolment to end of study period.

OTHER OUTCOMES:
Exploratory outcome: Maternal and perinatal adverse conditions | From time of enrolment to end of study period (6 weeks postpartum).
  maternal outcomes (maternal mortality, eclampsia, stroke, cortical blindness, retinal detachment, pulmonary edema, acute kidney injury, liver capsule hematoma or rupture, placental abruptions, post-partum hemorrhage, raised liver enzymes, low platelets, admission to intensive care unit, intubation and mechanical ventilation) and offspring outcomes (stillbirth, gestational age at delivery, birthweight, small for gestational age, neonatal mortality, neonatal seizures, admission to neonatal unit, and respiratory support)
Exploratory outcome: Efficacy as defined by proportion of blood pressure readings within guideline readings | From time of enrolment to end of study period (6 weeks postpartum).
  Proportion of home SBP and DBP under control defined as SBP < 135 mm Hg and DBP < 85 mm Hg as per national guidelines
Exploratory outcome: Efficacy as defined by mean blood pressures | 2nd trimester (up to 24 weeks of gestation), 3rd trimester (up to 36 weeks gestation), post-partum (up to 6 weeks post-partum)
  Mean home SBP and DBP under control defined as SBP < 135 mm Hg and DBP < 85 mm Hg as per national guidelines per trimester
Exploratory outcome: Process outcomes | 2nd trimester (up to 24 weeks of gestation), 3rd trimester (up to 36 weeks gestation), post-partum (up to 6 weeks post-partum)
  Number of alerts, phone calls, and technical issues between patients to health team
Exploratory outcome: Anti-hypertensive medications changes | 2nd trimester (up to 24 weeks of gestation), 3rd trimester (up to 36 weeks gestation), post-partum (up to 6 weeks post-partum)
  Number of changes to anti-hypertensive medications prescribed during the study period.
Exploratory outcome: Type of medications prescribed | 2nd trimester (up to 24 weeks of gestation), 3rd trimester (up to 36 weeks gestation), post-partum (up to 6 weeks post-partum)
  Type of anti-hypertensives that prescribed to patients during the study period
Exploratory outcome: Dose of medications prescribed | 2nd trimester (up to 24 weeks of gestation), 3rd trimester (up to 36 weeks gestation), post-partum (up to 6 weeks post-partum)
  Dose of anti-hypertensive medications that are prescribed to patients during the study period
Exploratory outcome: Fidelity to interventions | 2nd trimester (up to 24 weeks of gestation), 3rd trimester (up to 36 weeks gestation), post-partum (up to 6 weeks post-partum)
  Adherence to HBPT measured by proportion of: completed 7-day home BP series, anti-hypertensive titration instructions followed correctly and number of study visits attended.
Exploratory outcome: Health care utilization | From time of enrolment to end of study period (6 weeks postpartum).
  Number of unscheduled prenatal, emergency room or urgent care visits antenatal and post-partum, in person clinical assessments, and tele-health visits

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No